CLINICAL TRIAL: NCT02692040
Title: A Randomised, Placebo Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Gut Hormone Analogue G3215 in Adult Subjects
Brief Title: Study of the Gut Hormone Analogue G3215 in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/G3215/01
Record Dates: First submitted 2016-01-18; First posted 2016-02-25 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: obesity; diabetes mellitus; glucagon-like peptide-1
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (19):
- 12-24 mg (B1) dose of G3215 (Experimental): G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses to a max of 24 mg.
  Interventions: Drug: G3215
- 6-10 mg (B2) dose of G3215 (Experimental): G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses to a max of 10 mg.
  Interventions: Drug: G3215
- 5-16 mg (B3) dose of G3215 (Experimental): G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses to a max of 16 mg.
  Interventions: Drug: G3215
- 3.2mg (C) infusion pump dose of G3215 (Experimental): G3215 subcutaneous infusion over a 4 day treatment period at escalating doses to a max of 3.2 mg (with either the first or last day administering infusion of placebo [saline]).
  Interventions: Drug: G3215; Drug: Placebo
- Placebo (B) - saline (Placebo Comparator): 5 subcutaneous injections of 0.9% saline, over a 4 week treatment period
  Interventions: Drug: Placebo
- Placebo (A) - saline (Placebo Comparator): Single subcutaneous injection of 0.9% saline
  Interventions: Drug: Placebo
- 0.1 mg dose G3215 (A1) (Experimental): 0.1 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 0.5 mg dose G3215 (A1) (Experimental): 0.5 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 1.5 mg dose G3215 (A1) (Experimental): 1.5 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 4 mg dose G3215 (A2) with varied formulation (Experimental): 4 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 4 mg dose G3215 (A3) with varied formulation (Experimental): 4 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 4 mg dose G3215 (A4) with varied formulation (Experimental): 4 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 4 mg dose G3215 (A5) with varied formulation (Experimental): 4 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 8 mg dose G3215 (A7) (Experimental): 8 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 10 mg dose G3215 (A6) (Experimental): 10 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 12 mg dose G3215 (A8) (Experimental): 12 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 16 mg dose G3215 (A9) (Experimental): 16 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 32 mg dose G3215 (A10) (Experimental): 32 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215
- 48 mg dose G3215 (A11) (Experimental): 48 mg G3215 single dose, subcutaneous injection
  Interventions: Drug: G3215

INTERVENTIONS:
Drug: G3215 — Gut hormone analogue
  Arms: 0.1 mg dose G3215 (A1); 0.5 mg dose G3215 (A1); 1.5 mg dose G3215 (A1); 10 mg dose G3215 (A6); 12 mg dose G3215 (A8); 12-24 mg (B1) dose of G3215; 16 mg dose G3215 (A9); 3.2mg (C) infusion pump dose of G3215; 32 mg dose G3215 (A10); 4 mg dose G3215 (A2) with varied formulation; 4 mg dose G3215 (A3) with varied formulation; 4 mg dose G3215 (A4) with varied formulation; 4 mg dose G3215 (A5) with varied formulation; 48 mg dose G3215 (A11); 5-16 mg (B3) dose of G3215; 6-10 mg (B2) dose of G3215; 8 mg dose G3215 (A7)
Drug: Placebo — 0.9% saline
  Other Names: Saline
  Arms: 3.2mg (C) infusion pump dose of G3215; Placebo (A) - saline; Placebo (B) - saline

SUMMARY:
A randomised, placebo controlled Phase I study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of G3215 in adult subjects.

DETAILED DESCRIPTION:
Objectives:

Primary Objective

* To investigate the safety and tolerability of single doses of G3215 in overweight but otherwise healthy male subjects.
* To investigate the safety and tolerability of multiple doses of G3215 in overweight male subjects with mild stable Type 2 diabetes or prediabetes.

Secondary Objectives • To assess the pharmacokinetic (PK) profile of single and multiple ascending doses of G3215 in overweight but otherwise healthy male subjects or overweight / obese male subjects with mild stable Type 2 diabetes or prediabetes.

Exploratory Objective

• To investigate the effects of multiple doses of G3215 on food consumption, body weight, enteropancreatic hormone changes and glucose tolerance in overweight male subjects with mild Type 2 diabetes or prediabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18 to 60 years inclusive with body mass index (BMI) between 25.0 and 35.0 kg/m2 inclusive;
2. Subjects who are otherwise healthy enough to participate, as determined by pre-study medical history, physical examination and 12 lead ECG;
3. Subjects whose clinical laboratory test results are either within the normal range or if outside this range the abnormalities are judged to be not clinically relevant and are acceptable to the Investigator;
4. Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening;
5. Subjects who are negative for drugs of abuse and alcohol tests at screening and admissions;
6. Subjects who are non-smokers for at least 3 months preceding screening;
7. Subjects who agree to use medically acceptable methods of contraception for at least 3 months after study drug administration;
8. Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

1. Subjects who do not conform to the above inclusion criteria;
2. Subjects who have a clinically relevant history or presence of gastrointestinal (especially associated with vomiting), respiratory, renal, hepatic, haematological, lymphatic, neurological (especially if associated with balance disorders or vomiting e.g. migraine or labyrinthitis), cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders;
3. Subjects who have a clinically relevant surgical history;
4. Subjects who are currently taking thiazolidinediones, dipeptidyl peptidase IV inhibitors ('gliptins'), glucagon-like peptide-1 (GLP-1) analogues, sodium-glucose co-transporter (SGLT-2) inhibitors, and insulin;
5. Subjects who have a history of relevant and severe atopy e.g. asthma, angioedema requiring emergency treatment, severe hayfever requiring regular treatment, severe eczema requiring regular treatment;
6. Subjects who have a history of relevant drug hypersensitivity;
7. Subjects who have a history of alcohol abuse or alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria within the last two years;
8. Subjects who have a history of drug or substance abuse according to DSM-IV criteria within the last 2 years;
9. Subjects who have a history of clinically significant migraine as judged by the Investigator. Subjects can be included if they have not had a migraine for the last 3 years;
10. Subjects with a history of pancreatitis or pancreatic cancer;
11. Subjects who consume more than 21 units of alcohol a week (unit = 1 glass of wine (125 mL) = 1 measure of spirits = ½ pint of beer);
12. Subjects who have a significant infection or known inflammatory process on screening;
13. Subjects who have acute gastrointestinal symptoms at the time of screening or admission (e.g. nausea, vomiting, diarrhoea, heartburn);
14. Subjects who have an acute infection such as influenza at the time of screening or admission;
15. Subjects who have used prescription drugs within 2 weeks of first dosing. For Part B, patients are allowed; monotherapy with sulphonylureas, or metformin. In addition patients in Part B are allowed to take hypolipidaemic and/or antihypertensive treatments, provided that the doses have not been altered within the 4 weeks prior to entering the study. Other medications may be allowed if the Investigator and Sponsor both agree that they will not affect the outcome of the study or the safety of the subject.
16. Subjects who have used over the counter medication excluding routine vitamins and paracetamol but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 7 days of first dosing, unless agreed as not clinically relevant by the Principal Investigator and Sponsor;
17. Subjects who have donated blood within 3 months prior to screening; Subjects who have donated plasma within the 7 days prior to screening; Subjects who have donated platelets within the 6 weeks prior to screening
18. Subjects who have used any investigational drug in any clinical trial within 3 months of their first admission date;
19. Subjects who have received the last dose of investigational drug greater than 3 months ago but who are on extended follow-up;
20. Subjects who have previously received G3215;
21. Subjects who are vegans or have any dietary restrictions;
22. Subjects who cannot communicate reliably with the Investigator;
23. Subjects who are unlikely to co-operate with the requirements of the study;
24. History or evidence of abnormal eating behaviour, as observed through the Dutch Eating Behaviour (DEBQ) and SCOFF (Sick, Control, One Stone, Fat, Food) questionnaires at screening.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, PhD MRCS, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited by Covance Clinical Research Unit, Leeds, UK
Groups:
- Placebo (A) - Saline: 0.9% saline single subcutaneous injection
  Placebo: 0.9% saline
- G3215 Single Ascending Dose (A1): Sequential cross-over group received either Saline or 0.1 mg dose G3215 (A1) single dose, subcutaneous injection in the first treatment period; Saline or 0.5 mg dose G3215 single dose, subcutaneous injection in the second period, Saline or 1.5 mg dose G3215 single dose, subcutaneous injection in the third treatment period. Treatment periods were 12-15 days apart.
- Placebo (B) - Saline: 0.9% saline multiple subcutaneous injection:
  5 injections over a 4 week treatment period
  Placebo: 0.9% saline
- 12-24 mg (B1) Dose of G3215: G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses to a max of 24 mg.
  G3215: Gut hormone analogue
- 6-10 mg (B2) Dose of G3215: G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses to a max of 10 mg.
  G3215: Gut hormone analogue
- 5-16 mg (B3) Dose of G3215: G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses to a max of 16 mg.
  G3215: Gut hormone analogue
Period: Overall Study
Arm/Group | Placebo (A) - Saline | G3215 Single Ascending Dose (A1) | 4 mg Dose G3215 (A2) With Varied Formulation | 4 mg Dose G3215 (A3) With Varied Formulation | 4 mg Dose G3215 (A4) With Varied Formulation | 4 mg Dose G3215 (A5) With Varied Formulation | 8 mg Dose G3215 (A7) | 10 mg Dose G3215 (A6) | 12 mg Dose G3215 (A8) | 16 mg Dose G3215 (A9) | 32 mg Dose G3215 (A10) | 48 mg Dose G3215 (A11) | Placebo (B) - Saline | 12-24 mg (B1) Dose of G3215 | 6-10 mg (B2) Dose of G3215 | 5-16 mg (B3) Dose of G3215 | 3.2mg (C) Infusion Pump Dose of G3215
Started | 10 | 4 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 4
Completed | 10 | 4 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 5 | 3 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 90 male subjects entered the study and were randomised to treatment across Part A Single-dose (62 participants), Part B Multiple Ascending-dose (24 participants), and Part C (4 participants). In cohort 1 of Part A (SAD A1), 4 subjects received study drug (G3215 or saline) in 3 treatment periods; all other subjects in part A (A2-A11) received only a single dose.
Groups:
- Placebo (A2-A11) - Saline: Single subcutaneous injection of 0.9% saline
- 4 mg Dose G3215 (A2); 4 mg Dose G3215 (A3); 4 mg Dose G3215 (A4); 4 mg Dose G3215 (A5): 4 mg G3215 single dose, subcutaneous injection
- Placebo (B) - Saline: 0.9% saline multiple subcutaneous injection
  5 injections over a 4 week treatment period
  Placebo: 0.9% saline
- Total: Total of all reporting groups
Arm/Group | Placebo (A2-A11) - Saline | G3215 Single Ascending Dose (A1) | 4 mg Dose G3215 (A2) | 4 mg Dose G3215 (A3) | 4 mg Dose G3215 (A4) | 4 mg Dose G3215 (A5) | 8 mg Dose G3215 (A7) | 10 mg Dose G3215 (A6) | 12 mg Dose G3215 (A8) | 16 mg Dose G3215 (A9) | 32 mg Dose G3215 (A10) | 48 mg Dose G3215 (A11) | Placebo (B) - Saline | 12-24 mg (B1) Dose of G3215 | 6-10 mg (B2) Dose of G3215 | 5-16 mg (B3) Dose of G3215 | 3.2mg (C) Infusion Pump Dose of G3215 | Total
Number analyzed (Participants) | 10 | 4 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 4 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (16.2) | 47 (14.0) | 39 (7.3) | 40 (8.8) | 38 (10.1) | 47 (14.3) | 30 (15.2) | 48 (7.9) | 33 (12.8) | 45 (9.0) | 39 (11.7) | 49 (10.9) | 47 (8.7) | 45 (4.3) | 47 (13.7) | 45 (14.0) | 48 (16.3) | 42.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 4 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 4 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 4 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 4 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 4 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 4 | 98
Body Weight (kg) [Mean (Standard Deviation); unit: kg] | 88.9 (10.20) | 89.2 (7.75) | 83.7 (7.98) | 99.6 (10.72) | 94.6 (7.00) | 92.2 (9.34) | 92.3 (8.46) | 92.1 (9.48) | 92.4 (8.32) | 96.3 (16.36) | 89.3 (5.16) | 85.9 (14.88) | 88.3 (10.42) | 90.2 (3.08) | 92.1 (13.72) | 93.6 (13.51) | 87.9 (5.68) | 90.9 (9.9)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (2.51) | 29.1 (1.80) | 27.4 (1.94) | 29.8 (2.97) | 28.5 (2.46) | 29.5 (2.24) | 30.0 (2.98) | 29.3 (3.45) | 28.2 (2.50) | 29.7 (4.31) | 28.8 (1.78) | 28.0 (3.38) | 28.6 (3.72) | 29.0 (1.76) | 29.4 (3.94) | 29.5 (3.40) | 29.0 (1.48) | 28.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) [Safety and Tolerability]
Description: As assessed by reporting of adverse events, vital signs, physical examination, clinical laboratory safety assessments, and ECG parameters.
  Possibly or definitely related to study drug
Time Frame: up to 28 days after dosing
Measure: Count of Participants; unit: Participants
Groups:
- 4 mg Dose G3215 (A2); 4 mg Dose G3215 (A3); 4 mg Dose G3215 (A4); 4 mg Dose G3215 (A5): 4 mg G3215 single dose, subcutaneous injection
  G3215: Gut hormone analogue
- 5mg G3215 (B); 6 mg G3215 (B): G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses
  G3215: Gut hormone analogue
- 7 mg G3215 (B); 8 mg G3215 (B); 10 mg G3215 (B); 12 mg G3215 (B); 16 mg G3215 (B); 20 mg G3215 (B); 24 mg G3215 (B): G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses.
  G3215: Gut hormone analogue
- Placebo (C): Placebo: 0.9% saline
- 0.6 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 0.6 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 0.7 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 0.7 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 0.8 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 0.8 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 1 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 1 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 1.1 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 1.1 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 1.4 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 1.4 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 1.5 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 1.5 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 1.8 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 1.8 mg over 24h treatment period.
  G3215: Gut hormone analogue
- 2.2 mg/24h (C) Infusion Pump Dose of G3215: G3215 subcutaneous infusion of 2.2 mg over 24h treatment period.
  G3215: Gut hormone analogue
Arm/Group | Placebo (A) - Saline | 0.1 mg Dose G3215 (A1) | 0.5 mg Dose G3215 (A1) | 1.5 mg Dose G3215 (A1) | 4 mg Dose G3215 (A2) | 4 mg Dose G3215 (A3) | 4 mg Dose G3215 (A4) | 4 mg Dose G3215 (A5) | 8 mg Dose G3215 (A7) | 10 mg Dose G3215 (A6) | 12 mg Dose G3215 (A8) | 16 mg Dose G3215 (A9) | 32 mg Dose G3215 (A10) | 48 mg Dose G3215 (A11) | Placebo (B) - Saline | 5mg G3215 (B) | 6 mg G3215 (B) | 7 mg G3215 (B) | 8 mg G3215 (B) | 10 mg G3215 (B) | 12 mg G3215 (B) | 16 mg G3215 (B) | 20 mg G3215 (B) | 24 mg G3215 (B) | Placebo (C) | 0.6 mg/24h (C) Infusion Pump Dose of G3215 | 0.7 mg/24h (C) Infusion Pump Dose of G3215 | 0.8 mg/24h (C) Infusion Pump Dose of G3215 | 1 mg/24h (C) Infusion Pump Dose of G3215 | 1.1 mg/24h (C) Infusion Pump Dose of G3215 | 1.4 mg/24h (C) Infusion Pump Dose of G3215 | 1.5 mg/24h (C) Infusion Pump Dose of G3215 | 1.8 mg/24h (C) Infusion Pump Dose of G3215 | 2.2 mg/24h (C) Infusion Pump Dose of G3215
Number analyzed (Participants) | 13 | 3 | 3 | 3 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 8 | 1 | 7 | 3 | 6 | 4 | 1 | 2 | 1 | 1 | 1 | 1 | 3 | 1 | 1
Participants | 2 | 0 | 0 | 3 | 4 | 4 | 2 | 4 | 4 | 5 | 5 | 4 | 5 | 5 | 2 | 5 | 6 | 5 | 6 | 7 | 0 | 4 | 3 | 6 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 1 | 1

2. Secondary Outcome: Body Weight (Percentage Change From Baseline)
Description: Summary of Time-Matched % Change from Baseline in Body Weight (AM Baseline = Day 1 AM; PM Baseline = Day -1 PM
Time Frame: up to day 4 (am) for Part A, day 31 (pm) for Part B and day 5 (am) for Part C
Population: Completers
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Placebo (A) - Saline; Placebo (B) - Saline: 0.9% saline
  Placebo: 0.9% saline
- Infusion Pump Dose of G3215 (C): G3215 subcutaneous infusion over a 4 day treatment period at escalating doses to a max of 3.2 mg (with either the first or last day administering infusion of placebo [saline]).
  G3215: Gut hormone analogue
  Placebo: 0.9% saline
- Placebo (Part C): Placebo infusion received on day 4 of infusion pump study
Arm/Group | Placebo (A) - Saline | 0.1 mg Dose G3215 (A1) | 0.5 mg Dose G3215 (A1) | 1.5 mg Dose G3215 (A1) | 4 mg Dose G3215 (A2) | 4 mg Dose G3215 (A3) | 4 mg Dose G3215 (A4) | 4 mg Dose G3215 (A5) | 8 mg Dose G3215 (A7) | 10 mg Dose G3215 (A6) | 12 mg Dose G3215 (A8) | 16 mg Dose G3215 (A9) | 32 mg Dose G3215 (A10) | 48 mg Dose G3215 (A11) | Placebo (B) - Saline | 12-24 mg (B1) Dose of G3215 | 6-10 mg (B2) Dose of G3215 | 5-16 mg (B3) Dose of G3215 | Infusion Pump Dose of G3215 (C) | Placebo (Part C)
Number analyzed (Participants) | 13 | 3 | 3 | 3 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 5 | 5 | 3 | 5 | 4 | 2 | 2
Percentage change | 0.1 (0.97) | 0.2 (0.47) | 0.8 (0.15) | 0.1 (0.42) | 0.9 (0.68) | 0.2 (0.49) | -0.7 (0.29) | 0.4 (0.7) | -0.7 (0.73) | -1.4 (0.44) | -0.1 (0.53) | -0.1 (0.51) | -1.7 (1.16) | -0.9 (0.74) | -1.4 (1.26) | -3.7 (2.58) | -5.3 (3.79) | -4.5 (1.72) | -3.2 (0) | -3.0 (0)

ADVERSE EVENTS:
Time Frame: Up to 21 weeks from participant start date
Description: The safety evaluation will include blood pressure, pulse rate, ECG parameters, clinical laboratory tests (haematology, serum biochemistry, coagulation, urinalysis and urine microscopy).
Groups:
- Placebo (A) - Saline: 0.9% saline, single dose, subcutaneous injection
  Placebo: 0.9% saline
- Placebo (B) - Saline: 0.9% saline, multiple subcutaneous injections 5 injections over a 4 week treatment period
  Placebo: 0.9% saline
- 5 mg G3215 (B); 6 mg G3215 (B); 7 mg G3215 (B); 8 mg G3215 (B); 10 mg G3215 (B); 12 mg G3215 (B); 16 mg G3215 (B); 20 mg G3215 (B); 24 mg G3215 (B): G3215 multiple dose, subcutaneous injection:
  5 doses over a 4 week treatment period at escalating doses.
  G3215: Gut hormone analogue
- Placebo (C): Placebo: 0.9% saline subcutaneous infusion over a 24 hour treatment period
- 0.6 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 0.6 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 0.7 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 0.7 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 0.8 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 0.8 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 1 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 1 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 1.1 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 1.1 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 1.4 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 1.4 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 1.5 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 1.5 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 1.8 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 1.8 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
- 2.2 mg/24h (C) Infusion Rate Pump of G3215: G3215 subcutaneous infusion of 2.2 mg over a 24 hour treatment period
  G3215: Gut hormone analogue
Arm/Group | Placebo (A) - Saline | 0.1 mg Dose G3215 (A1) | 0.5 mg Dose G3215 (A1) | 1.5 mg Dose G3215 (A1) | 4 mg Dose G3215 (A2) | 4 mg Dose G3215 (A3) | 4 mg Dose G3215 (A4) | 4 mg Dose G3215 (A5) | 8 mg Dose G3215 (A7) | 10 mg Dose G3215 (A6) | 12 mg Dose G3215 (A8) | 16 mg Dose G3215 (A9) | 32 mg Dose G3215 (A10) | 48 mg Dose G3215 (A11) | Placebo (B) - Saline | 5 mg G3215 (B) | 6 mg G3215 (B) | 7 mg G3215 (B) | 8 mg G3215 (B) | 10 mg G3215 (B) | 12 mg G3215 (B) | 16 mg G3215 (B) | 20 mg G3215 (B) | 24 mg G3215 (B) | Placebo (C) | 0.6 mg/24h (C) Infusion Rate Pump of G3215 | 0.7 mg/24h (C) Infusion Rate Pump of G3215 | 0.8 mg/24h (C) Infusion Rate Pump of G3215 | 1 mg/24h (C) Infusion Rate Pump of G3215 | 1.1 mg/24h (C) Infusion Rate Pump of G3215 | 1.4 mg/24h (C) Infusion Rate Pump of G3215 | 1.5 mg/24h (C) Infusion Rate Pump of G3215 | 1.8 mg/24h (C) Infusion Rate Pump of G3215 | 2.2 mg/24h (C) Infusion Rate Pump of G3215
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/3 | 0/3 | 0/3 | 0/5 | 0/5 | 1/4 | 0/5 | 0/5 | 0/5 | 0/5 | 0/4 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/1 | 0/7 | 3/3 | 6/6 | 4/4 | 1/1 | 2/2 | 1/1 | 1/1 | 1/1 | 1/1 | 3/3 | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3 | 0/3 | 0/3 | 0/5 | 0/5 | 1/4 | 0/5 | 0/5 | 0/5 | 0/5 | 0/4 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/1 | 0/7 | 0/3 | 0/6 | 0/4 | 0/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 5/13 | 1/3 | 3/3 | 3/3 | 5/5 | 4/5 | 4/4 | 4/5 | 4/5 | 5/5 | 5/5 | 4/4 | 5/5 | 5/5 | 5/6 | 5/6 | 6/6 | 6/6 | 6/6 | 7/8 | 0/1 | 5/7 | 3/3 | 6/6 | 1/4 | 1/1 | 2/2 | 0/1 | 1/1 | 1/1 | 1/1 | 2/3 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (A) - Saline (N=13) | 0.1 mg Dose G3215 (A1) (N=3) | 0.5 mg Dose G3215 (A1) (N=3) | 1.5 mg Dose G3215 (A1) (N=3) | 4 mg Dose G3215 (A2) (N=5) | 4 mg Dose G3215 (A3) (N=5) | 4 mg Dose G3215 (A4) (N=4) | 4 mg Dose G3215 (A5) (N=5) | 8 mg Dose G3215 (A7) (N=5) | 10 mg Dose G3215 (A6) (N=5) | 12 mg Dose G3215 (A8) (N=5) | 16 mg Dose G3215 (A9) (N=4) | 32 mg Dose G3215 (A10) (N=5) | 48 mg Dose G3215 (A11) (N=5) | Placebo (B) - Saline (N=6) | 5 mg G3215 (B) (N=6) | 6 mg G3215 (B) (N=6) | 7 mg G3215 (B) (N=6) | 8 mg G3215 (B) (N=6) | 10 mg G3215 (B) (N=8) | 12 mg G3215 (B) (N=1) | 16 mg G3215 (B) (N=7) | 20 mg G3215 (B) (N=3) | 24 mg G3215 (B) (N=6) | Placebo (C) (N=4) | 0.6 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 0.7 mg/24h (C) Infusion Rate Pump of G3215 (N=2) | 0.8 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1.1 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1.4 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1.5 mg/24h (C) Infusion Rate Pump of G3215 (N=3) | 1.8 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 2.2 mg/24h (C) Infusion Rate Pump of G3215 (N=1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (A) - Saline (N=13) | 0.1 mg Dose G3215 (A1) (N=3) | 0.5 mg Dose G3215 (A1) (N=3) | 1.5 mg Dose G3215 (A1) (N=3) | 4 mg Dose G3215 (A2) (N=5) | 4 mg Dose G3215 (A3) (N=5) | 4 mg Dose G3215 (A4) (N=4) | 4 mg Dose G3215 (A5) (N=5) | 8 mg Dose G3215 (A7) (N=5) | 10 mg Dose G3215 (A6) (N=5) | 12 mg Dose G3215 (A8) (N=5) | 16 mg Dose G3215 (A9) (N=4) | 32 mg Dose G3215 (A10) (N=5) | 48 mg Dose G3215 (A11) (N=5) | Placebo (B) - Saline (N=6) | 5 mg G3215 (B) (N=6) | 6 mg G3215 (B) (N=6) | 7 mg G3215 (B) (N=6) | 8 mg G3215 (B) (N=6) | 10 mg G3215 (B) (N=8) | 12 mg G3215 (B) (N=1) | 16 mg G3215 (B) (N=7) | 20 mg G3215 (B) (N=3) | 24 mg G3215 (B) (N=6) | Placebo (C) (N=4) | 0.6 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 0.7 mg/24h (C) Infusion Rate Pump of G3215 (N=2) | 0.8 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1.1 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1.4 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 1.5 mg/24h (C) Infusion Rate Pump of G3215 (N=3) | 1.8 mg/24h (C) Infusion Rate Pump of G3215 (N=1) | 2.2 mg/24h (C) Infusion Rate Pump of G3215 (N=1)
Injection Site mass (General disorders) | 0 | 0 | 0 | 3 (3) | 4 (4) | 4 (4) | 2 (2) | 0 | 2 (2) | 3 (3) | 5 (5) | 4 (5) | 4 (4) | 5 (5) | 0 | 0 | 4 (14) | 3 (7) | 2 (3) | 4 (9) | 0 | 3 (5) | 2 (4) | 4 (17) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 0 | 0 | 2 (3) | 2 (2) | 1 (1) | 4 (7) | 0 | 2 (3) | 2 (4) | 6 (13) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (5) | 0 | 0 | 1 (1) | 1 (4) | 0 | 0 | 0 | 1 (1) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (3) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 3 (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 | 0 | 2 (5) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 | 3 (3) | 5 (10) | 2 (3) | 3 (3) | 6 (15) | 3 (6) | 5 (5) | 2 (3) | 0 | 1 (1) | 2 (2) | 3 (11) | 0 | 1 (2) | 2 (2) | 0 | 1 (1) | 1 (2) | 1 (6) | 2 (4) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 2 (2) | 0 | 0 | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 4 (6) | 3 (4) | 3 (3) | 5 (9) | 0 | 0 | 0 | 4 (9) | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 1 (3) | 2 (2) | 1 (2) | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 1 (1) | 3 (3) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (2) | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 (2) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 2 (2) | 0 | 0 | 1 (1) | 1 (2) | 2 (5) | 0 | 2 (2) | 0 | 2 (3) | 1 (2) | 0 | 0 | 1 (1) | 2 (6) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 | 0 | 0 | 3 (4) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (4) | 0 | 0 | 2 (2) | 5 (5) | 1 (1) | 5 (5) | 5 (6) | 3 (3) | 4 (5) | 3 (3) | 0 | 0 | 0 | 3 (5) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (3)
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Instillation site warmth (General disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 (0) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT02692040/Prot_SAP_000.pdf